CLINICAL TRIAL: NCT05159232
Title: Length of Hospital Stay in Laparoscopic Transabdominal Preperitoneal Vs. Open Mesh Repair in Inguinal Hernia: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memon Medical Institute (Other)
Collaborators: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, salma khan, Assistant Prof Surgery, Khyber Medical College, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IREB#194-SUR-2018
Record Dates: First submitted 2021-11-30; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Length of Stay

STUDY DESIGN:
Intervention Model Description: non-probability consecutive sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic trans abdominal preperitoneal repair (Active Comparator): length of hospital stay
  Interventions: Procedure: hospital stay
- open mesh repair of inguinal hernia (Active Comparator): length of hospital stay
  Interventions: Procedure: hospital stay

INTERVENTIONS:
Procedure: hospital stay — hospital stay in in inguinal hernia repair

SUMMARY:
To compare the mean length of hospital stay in laparoscopic trans abdominal preperitoneal repair versus open mesh repair in patients undergoing inguinal hernia repair with mesh.

DETAILED DESCRIPTION:
A total of 334 patients of male gender with Inguinal hernias of any side and ASA score I and II were included in the study. History of Immunosuppression, associated with other abdominal hernias and recurrent hernia were excluded. 167 patients were in Group A or laparoscopic trans abdominal preperitoneal repair group while 167 patients were in Group B or open mesh repair. Data regarding length of hospital stay from both groups was recorded by researcher himself on especially designed proforma.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-60 years

  * Inguinal hernias of any side as per operational definition
  * ASA score I and II

Exclusion Criteria:

* • H/o Immunosuppression

  * Associated with other abdominal hernias
  * H/o recurrent hernia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — all male patients
Enrollment: 334 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Duration of hospitals stay | 1-2 days
  hospital stay in hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salma khan, FCPS, Principal Investigator — rehman Medical Institute hospital
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No